CLINICAL TRIAL: NCT06432660
Title: Prospective Registry of Ocular Melanoma Eye Plaque brachyTherapy Patients (PROMPT)
Brief Title: Eye Plaque Brachytherapy for Ocular Melanoma
Acronym: PROMPT
Status: Active, not recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00115893
Record Dates: First submitted 2024-05-23; First posted 2024-05-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Ocular Melanoma
Keywords: eye plaque brachytherapy
MeSH Terms: conditions — Uveal Melanoma | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ocular Melanoma: Patients 18 years of age or older with unilateral primary choroidal melanoma
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Information about radiation therapy via eye plaque brachytherapy and follow up

SUMMARY:
This prospective registry study will evaluate doses utilized in eye plaque brachytherapy for the treatment of ocular melanoma and their associated outcomes. The goal of this study is to evaluate if lower doses of radiation can maintain high local control rates while minimizing the toxicities related to radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older with unilateral primary choroidal melanoma
* Patients with diagnosis of small or medium ocular melanomas amenable to plaque brachytherapy (as determined by treating ocular oncologist). Typically this would include tumors with apical height ≤10mm and basal diameter ≤16mm (small and medium tumors per COMS (Collaborative Ocular Melanoma Study)
* Patients with no clinical evidence of metastatic disease as confirmed by negative staging imaging (CT, MRI, and/or ultrasound)
* Patients with best-corrected visual acuity in the fellow eye of 20/200 or better
* Patients must be treated with IsoAid Eye Physics eye plaques

Exclusion Criteria:

* Patients whose tumors are circumferential around the optic disc and cannot be adequately covered by the prescription dose are ineligible.
* Similarly, patients with extrascleral tumor extension detected during echography or clinical exam, diffuse, ring or multifocal tumors that cannot be encompassed in a single episcleral plaque or tumors judged to be predominantly ciliary body or iris melanoma will be considered ineligible
* Previous treatment for ocular melanoma in either eye or treatment of any condition secondary to the tumor are ineligible.
* Patients with a history of other primary or metastatic cancers are not eligible, except for non-melanotic skin cancers
* Patients with extraocular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients seen at the Duke Eye Center and/or Duke Department of Radiation Oncology who meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2024-07-03 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with no disease recurrence within the radiation therapy field. | 5 years
  Number of disease free participants expressed as a percentage of the total number of participants enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Dianda Ayala-Peacock, MD, Principal Investigator — Duke University Health System (DUHS)
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meltsner SG, Rodrigues A, Materin MA, Kirsch DG, Craciunescu O. Transitioning from a COMS-based plaque brachytherapy program to using eye physics plaques and plaque simulator treatment planning system: A single institutional experience. J Appl Clin Med Phys. 2023 May;24(5):e13902. doi: 10.1002/acm2.13902. Epub 2023 Jan 13. PMID 36637797